CLINICAL TRIAL: NCT06402734
Title: Effects of Gluten-Free Diet on Nutritional Status and Inflammation Parameters in Adult Celiac Patients
Brief Title: Effects of Gluten-Free Diet on Nutritional Status in Celiac Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Associate Professor, Hacettepe University
Other Study IDs: GO 18/760
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Celiac Disease
Keywords: celiac disease; inflammation; interferon-gamma; interleukin-15
MeSH Terms: conditions — Celiac Disease; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples were collected from all subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac Disease: Adult patients who were diagnosed with celiac disease were enrolled in the study.
  Interventions: Behavioral: Adherence to Gluten Free Diet
- Healthy Subjects: Healthy subjects with matching demographical characteristics to the celiac group were enrolled in the study.

INTERVENTIONS:
Behavioral: Adherence to Gluten Free Diet — Participants with a diagnosed celiac disease were following a gluten-free diet. Study observed the adherence to the gluten-free diet for 6 weeks.
  Groups: Celiac Disease

SUMMARY:
This study examined the impact of a gluten-free diet on nutritional status and inflammation markers in adult celiac patients compared to a control group. Twenty-six celiac patients and 26 healthy individuals participated. Interviews, dietary records, anthropometric measurements, and blood samples were collected. After six weeks, celiac patients showed improved adherence to the gluten-free diet and increased quality of life scores. While initial micronutrient intake was lower in celiac patients, it improved over the study period. However, there were no significant changes in inflammation markers.

DETAILED DESCRIPTION:
This study aimed to examine the effects of a gluten-free diet on the nutritional status, anthropometric measurements, and serum levels of interferon-gamma (IFN-γ) and interleukin-15 (IL-15) in adult celiac patients, comparing them with a control group. A total of 26 celiac patients aged 18-64 years and 26 healthy individuals as the control group were included. Face-to-face interviews were conducted to determine participants' general characteristics, dietary habits, and physical activity status. Additionally, a retrospective 24-hour dietary recall and food frequency questionnaire were administered to assess dietary intake. Anthropometric measurements and blood samples were collected during the interviews. Celiac patients received education about the gluten-free diet, and follow-up assessments were conducted six weeks later. At the beginning, 53.8% of celiac patients reported always/mostly adhering to the gluten-free diet, which increased to 100.0% after six weeks. The total quality of life scores significantly increased in celiac patients after six weeks. Initial serum IL-15 levels were similar between celiac and control groups, whereas serum IFN-γ levels were significantly higher in celiac patients compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 19 and 64 years old.
* Diagnosis of celiac disease.
* Willingness to participate in the study.
* Ability to adhere to the study protocol, including dietary restrictions and follow-up assessments.
* For the control group, individuals without celiac disease or any other significant health conditions.

Exclusion Criteria:

* Individuals following diets other than a gluten-free diet.
* Individuals adhering to a gluten-free diet for reasons other than celiac disease.
* Individuals with gastrointestinal diseases other than celiac disease.
* Individuals who have undergone gastrointestinal surgery.
* Individuals with mental illnesses.
* Cancer patients.
* Individuals positive for hepatitis B surface antigen or anti-hepatitis C virus antibody.
* Individuals using interferon and/or insulin.
* Pregnant or lactating women.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 26 individuals diagnosed with celiac disease, comprising 21 females and 5 males, aged between 18 and 64 years. Additionally, a healthy control group of 26 individuals, including 20 females and 6 males, without any known diseases, was included in the study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Serum interferon-gamma level | 6 weeks
  Serum interferon-gamma level was measured.
Serum interleukin-15 levels | 6 weeks
  Serum interleukin-15 level was measured.
Body weight | 6 weeks
  Body weight was measured using body composition analyzer device.
Lean body mass | 6 weeks
  Lean body mass was measured using body composition analyzer device.

SECONDARY OUTCOMES:
Total energy intake | 6 weeks
  Total energy intake was measured using food records.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Nutrition and Dietetics Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the ethical reasons participant data will not be shared.